CLINICAL TRIAL: NCT07048873
Title: Effect of Dexmedetomidine Versus Ketamine on Patients of Laryngeal Microsurgery: a Randomized Controlled Study
Brief Title: Dexmedetomidine Versus Ketamine on Laryngeal Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Ismail, Associate Professor of Anesthesia, Surgical ICU and pain management at Faculty of medicine Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-502-2023
Record Dates: First submitted 2024-05-05; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Microlaryngeal Surgery
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Sodium Chloride; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine (Experimental): 1.0mcg/kg of dexmedetomidineloading dose before induction then 0.5 mcg/kg/hr of infused till end of surgery
  Interventions: Drug: Dexmedetomidine
- Ketamine (Experimental): 0.25 mg/kg/hr ketamine infused till end of surgery
  Interventions: Drug: Ketamine
- Control (Active Comparator): saline before induction infusion till end of surgery
  Interventions: Drug: Saline (control group)

INTERVENTIONS:
Drug: Dexmedetomidine — IV dexmedetomidine
  Arms: Dexmedetomidine
Drug: Ketamine — IV ketamine
  Arms: Ketamine
Drug: Saline (control group) — no drugs
  Other Names: NO drugs
  Arms: Control

SUMMARY:
compare effect of IV dexmedetomidine and ketamine on pain score, perioperative hemodynamics and detect side effects of dexmedetomidine and ketamine.

DETAILED DESCRIPTION:
Microlaryngeal surgery is a common surgical procedure now a days which is associated with many complications such as postoperative pain, airway edema and persistent cough

. the study is to compare the effect of IV dexmedetomidine and ketamine on pain score, perioperative hemodynamics and to detect side effects of dexmedetomidine and ketamine.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years ASA I,II

Exclusion Criteria:

* CVdiseases as IHD and severe valvular disease.

  * allergy to ketamine or dexmedetomidine.
  * Patients refusal
  * Suspected difficult intubation more than 2 trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative sore throat | 30 minutes postoperative
  incidence of postoperative sore throat

SECONDARY OUTCOMES:
Ramsey sedation score | 1hour postoperative
  Ramsey sedation score RSS (1 to 6)
postoperative cough incidence | 1hour postoperative
  postoperative cough incidence
incidence of complications | 1hour postoperative
  incidence of complications
Heart Rate | 1hour postoperative
  Heart Rate
Mean Arterial Pressure | 1hour postoperative
  Mean Arterial Pressure
oxygen saturation | 1hour postoperative
  oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No